CLINICAL TRIAL: NCT02796885
Title: Characterisation of Adult-Onset Hypophosphatasia
Status: Completed | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: STH18683; 16/NW/0385 (Other: UK HRA REC); 202179 (Other: UK HRA IRAS)
Record Dates: First submitted 2016-05-04; First posted 2016-06-13 (Estimated); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Hypophosphatasia
MeSH Terms: conditions — Hypophosphatasia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum, plasma, urine, whole blood for DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Possible hypophosphatasia: Patients attending metabolic bone services, not previously know to have HPP, with biochemistry suggestive of HPP Will have TNSALP gene test, clinical assessment for possible features of HPP, bone turnover marker profile.
  Interventions: Other: no intervention - observational study
- Normal: Patients attending metabolic bone services, not previously know to have HPP, with normal HPP biochemistry Will have TNSALP gene test, clinical assessment for possible features of HPP, bone turnover marker profile.
  Interventions: Other: no intervention - observational study
- Known hypophosphatasia: Patients attending metabolic bone services or registered with RUDY database, known to have HPP Will have TNSALP gene test, clinical assessment for possible features of HPP, bone turnover marker profile.
  Interventions: Other: no intervention - observational study

INTERVENTIONS:
Other: no intervention - observational study

SUMMARY:
Hypophosphatasia (HPP) is an inherited condition which causes a defect in bone calcification, leading to weak bones. Early childhood forms are severe and easily recognised, and there is now a drug treatment which is very effective in children.

Adult forms are milder, often missed by doctors or confused with osteoporosis. This is important because the usual osteoporosis treatments may be harmful in HPP, and increase the risk of broken bones. One of the reasons it is missed is a lack of research describing the typical features of HPP, so doctors don't recognise the signs, and don't know when or how to test for it.

The aim of this study is to establish clear criteria (from clinical history, examination and blood tests) to identify people with HPP. The results will also determine if there should be a trial of drug treatment for adults with HPP.

DETAILED DESCRIPTION:
Hypophosphatasia (HPP) is a genetic disorder caused by mutation in the tissue-non-specific alkaline phosphatase gene (TNSALP). It causes impaired bone mineralisation, fractures, tooth loss, muscle weakness and possibly other adverse health outcomes.

The infantile-onset forms are severe, and were often fatal until the recent availability of a treatment (Asfotase Alfa, Alexion Pharma). The childhood-onset forms are less severe, and the adult-onset form is mild, and often unrecognised or misdiagnosed as osteoporosis.

The less severe forms of the disease are not well described, and because there has been no available treatment there has not been much research in adults. However, now that treatment is available there is a possibility of a clinical trial in adults.

Additionally, patients with hypophosphatasia are often not recognised, and are misdiagnosed as having osteoporosis. This is important because patients with hypophosphatasia are at risk of developing atypical femoral fractures if they are treated with usual osteoporosis medication (bisphosphonates).

A major contributor to the under-recognition of adult HPP is the lack of phenotypic description and biomarker definitions. The aim of this project is to identify the clinical and biochemical characteristics that identify HPP.

In preparation for this study reference ranges for the commonly used HPP biomarkers (ALP and PLP) have been established, and used to screen 2000 patients presenting to metabolic bone services in Sheffield and Oxford.

For this study, patients who have biochemistry suggestive of HPP (low ALP and high PLP), will undergo a detailed clinical assessment, with medical history, physical examination, bone biochemistry, targeted musculoskeletal imaging and HPP gene testing. Their results will be compared with a control group of metabolic bone clinic patients with normal ALP and PLP, and a group of patients with known gene-proven and clinically manifest HPP.

The results will establish clinical phenotype and biomarker criteria for HPP diagnosis, which could be incorporated into future pathways for patients presenting to metabolic bone clinics. This will improve the identification of HPP and prevent harm from incorrect treatment with bisphosphonates.

ELIGIBILITY:
Inclusion Criteria:

* As the groups described above
* Able and willing to participate in the study and provide written informed consent

Exclusion Criteria:

* Other conditions known to affect serum ALP and PLP (Coeliac disease, B12 deficiency, untreated hypothyroidism, Wilson's disease)
* Taking nutritional supplements containing vitamin B6
* Pregnant

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients attending metabolic bone services in Sheffield and Oxford, UK Patients with hypophosphatasia registered on the RUDY database.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
ALP and PLP | baseline cross-sectional
  predictive value of low ALP with high PLP for TNSALP mutation (ROC curve)

SECONDARY OUTCOMES:
ALP:PINP ratio | baseline cross-sectional
  predictive value of ALP:PINP ratio for TNSALP mutation (ROC curve)PP
prevalence of imaging-confirmed musculoskeletal pathology in patients with HPP | baseline cross-sectional
  History and clinical examination will be obtained to identify possible musculoskeletal pathology. Imaging (x-ray, ultrasound or MRI) will be obtained to determine the nature of the pathology. Will include arthritis, enthesopathy, tendonitis.
  Prevalence of musculoskeletal pathology in people with biochemistry suggestive of HPP and positive gene test will be compared with normal controls.
short physical function battery score | baseline cross-sectional
  physical function battery score in people with biochemistry suggestive of HPP and positive gene test (compared with normal controls)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Eastell, Principal Investigator — University of Sheffield
Locations (2):
- United Kingdom (2):
  - Nuffield Orthopaedic Research, Oxford
  - University of Sheffield, Sheffield